CLINICAL TRIAL: NCT02309593
Title: Post Market Clinical Follow-up Study Protocol for PROFEMUR® Xm Femoral Stems
Status: Terminated | Type: Observational
Why Stopped: PI change, hospital change and covid -19 caused lost-to-follow up of most of the subjects
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002A
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; painful hip dysplasia; rheumatoid arthritis; correction of functional deformity; revision procedures
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- PROFEMUR® Xm Femoral Stems: Single study group either previously implanted or will be implanted with the following combination of components: PROFEMUR® Xm Femoral Stems, with any type of Acetabular Shells.
  Interventions: Device: PROFEMUR® Xm Femoral Stems

INTERVENTIONS:
Device: PROFEMUR® Xm Femoral Stems — THA using PROFEMUR® Xm Femoral Stems
  Other Names: Primary hip replacement device

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) and resurfacing components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA and resurfacing devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject previously underwent / is a candidate for primary THA for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject has been previously implanted / is a candidate to be implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments
* Not previously implanted subject is able to undergo primary THA procedure

Previously implanted bilateral subjects can have both THAs enrolled in the study provided:

* the specified combination of components were implanted in both
* all other aspects of the Inclusion/Exclusion Criteria are satisfied
* enrollment does not exceed the subject count specified in the Clinical Trial Agreement
* the subject agrees to a second Informed Consent document specific to the second THA

Prospective enrollment of a previously unimplanted contralateral hip is permitted in this study provided:

* it occurs not more than two years after the index THA
* the specified combination of components is used
* all other aspects of the Inclusion/Exclusion Criteria are satisfied
* enrollment does not exceed the subject count specified in the Clinical Trial Agreement
* the subject agrees to a second Informed Consent document specific to the second THA

Exclusion Criteria:

* Subject is skeletally immature (less than 21 years of age) at time of primary THA surgery
* Subject is currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subject is unwilling to sign the Informed Consent document
* Subject has substance abuse issues
* Subject is incarcerated or has pending incarceration
* Subject is anticipated to require a contralateral THA less than 1 year after the index THA on the enrolled hip

In addition, not previously implanted subjects will be excluded if they meet any of the following criteria:

* Subject has any of the following contraindications at the time of implantation
* Overt infection
* Distant foci of infections (which may cause hematogenous spread to the implant site)
* Rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram
* Inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
* Neuropathic joints
* Hepatitis or HIV infection
* Neurological or musculoskeletal disease that may adversely affect gait or weight-bearing

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single study group either previously implanted or will be implanted with the following combination of components: PROFEMUR® Xm Femoral Stems, with any type of Acetabular Shells.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional outcomes (hip specific) | Previously implanted subjects: 6 months, 1, 3, 5, 7, and 10 years postoperatively beginning with first available visit; not previously implanted subjects: Pre-operative, 6 months, 1, 3, 5, 7, and 10 years postoperatively.
  To characterize total functional scores, as assessed by Oxford Hip Scores
Patient functional outcomes (quality of life) | Previously implanted subjects: 6 months, 1, 3, 5, 7, and 10 years postoperatively beginning with first available visit; not previously implanted subjects: Pre-operative, 6 months, 1, 3, 5, 7, and 10 years postoperatively.
  To characterize total functional scores, as assessed by EQ-5D-3L scores

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Jäger, MD, Principal Investigator — St. Marien-Hospital Mülheim
Locations (1):
- St. Marien-Hospital Mülheim, Klinik für Orthopädie, Unfall & Wiederherstellungschirurgie, Mülheim, Germany

IPD SHARING:
Plan to Share IPD: No